CLINICAL TRIAL: NCT00517595
Title: A Phase II Study of Pemetrexed and Gemcitabine Plus Bevacizumab as First Line Chemotherapy for Elderly Patients With Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Phase II Study Alimta and Gemzar + Avastin as First Line Chemotherapy for Elderly Patients With Stage IIIB/IV NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Eli Lilly and Company (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALJBNSCLC0602
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pemetrexed and Gemcitabine plus Bevacizumab — Bevacizumab 10 mg/kg will be given intravenously according to weight. Pemetrexed 500 mg/m^2 and gemcitabine 1500 mg/m^2 will be given intravenously according to weight and height. All agents are administered every 2 weeks.
  Other Names: Pemetrexed/Alimta; Gemcitabine/Gemzar; Bevacizumab/Avastin

SUMMARY:
The primary objective is to determine the progression free survival with pemetrexed, and gemcitabine plus bevacizumab as first-line chemotherapy in elderly patients with Stage IIIB/IV non-small cell lung cancer (NSCLC).

The secondary objectives are to determine the overall response rate; overall survival; chemotherapy induced toxicity profile of this combination; time to progression; and patient reported symptom burden.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Patient ≥ 65 years of age with ECOG of 0 to 1
* Patient must have histologically/cytologically confirmed Stage IIIB/IV NSCLC.
* Patient has measurable disease defined as at least 1 lesion that can be accurately measured in at least 1 dimension (by CT or MRI) & used to assess response as defined by RECIST criteria. Tumors within a previously irradiated field will be designated nontarget lesions.
* Patient has not received radiotherapy within 2 weeks(4 weeks required for brain metastases radiotherapy)of initial chemotherapy dosing for this study, and all acute toxicities due to prior radiotherapy have resolved prior to initial chemotherapy dosing.
* Patient has a negative serum pregnancy test or has undergone hysterectomy at time of enrollment.
* Greater than 12 weeks life expectancy.
* Patient has recovered from any recent surgery for at least 30 days & is free of active infection requiring antibiotics.
* Patient must be willing/able to discontinue use of NSAIDS prior to study drug dosing.
* Patient must be able to take folic acid, Vitamin B12, & dexamethasone per protocol.
* Patient must exhibit no greater than Grade 1 peripheral neuropathy.

Exclusion Criteria:

* Prior systemic or other concurrent chemo for metastatic NSCLC(Prior Tarceva is not allowed).Prior adjuvant chemo acceptable as long as > 12 months since completion and no prior pemetrexed, gemcitabine or bevacizumab.
* Lung carcinoma of squamous cell histology(mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is acceptable.Patients with extrathoracic-only squamous cell NSCLC are eligible.Patients with only peripheral lung lesions (of any NSCLC histology) will also be eligible(a peripheral lesion is defined as a lesion in which the epicenter of the tumor is ≤ 2 cm from the costal or diaphragmatic pleura in a three-dimensional orientation based on each lobe of the lung and is > 2 cm from the trachea, main, and lobar bronchi).
* Hemoptysis within 1 month prior to study enrollment
* Ongoing treatment with full-dose warfarin or its equivalent i.e., unfractionated and/or low molecular weight heparin.(Low dose warfarin 1 mg given for prophylaxis is allowed).
* Hypersensitivity to any component of Alimta, gemcitabine &/or bevacizumab, &/or cannot tolerate folic acid, corticosteroids or Vitamin B12 supplements.
* Currently/have recently taken long-acting NSAID (Ibuprofen ≤ 400 mg QID acceptable) or aspirin (>325mg/day) within 5 days of initial pemetrexed administration.
* Clinically significant pericardial/pleural effusion or ascites unless able to be drained before study entry.
* Presence of third space fluid which cannot be controlled by drainage.
* Core biopsy/other minor surgical procedure(excluding placement of a vascular access device)within 7 days prior to study enrollment.
* Active infection or fever ≥ 38.5°C within 3 days of first scheduled day of protocol treatment.
* Serious, non-healing wound, ulcer, or untreated bone fracture.
* NYHA Grade II or greater CHF
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 &/or diastolic blood pressure > 100mmHg on antihypertensive meds)
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* History of MI, CVA, TIA, or unstable angina within 6 months of study enrollment.
* Significant vascular disease (aortic aneurysm, aortic dissection or recent peripheral arterial thrombosis.)
* Symptomatic peripheral vascular disease
* Known bleeding diathesis or coagulopathy
* Presence of CNS(central nervous system) except for treated brain metastases. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging(MRI or CT)during the screening period.Anticonvulsants(stable dose)are allowed.Treatment for brain metastases may include whole brain radiotherapy(WBRT),radiosurgery(RS;Gamma Knife,LINAC,or equivalent)or a combination as deemed appropriate by the treating physician.Radiotherapy must be completed at least 4 weeks prior to study enrollment and all acute radiotherapy toxicities resolved.Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* A major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to enrollment.
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current prostate specific antigen of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry.
* Have received radiotherapy to more than 25% of their bone marrow.
* Receiving concurrent investigational therapy or has received investigational therapy within 30 days of the first scheduled day of protocol treatment
* Pregnant/lactating.
* Any other medical condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate/participate in the study, or interfere with interpretation of the results.
* History of allogeneic transplant.
* Known HIV infection or Hepatitis B or C.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnetta L Blakely, MD, Principal Investigator — Accelerated Community Oncology Research Network
Locations (10):
- United States (10):
  - Medical Oncology & Hematology, Waterbury, Connecticut
  - Augusta Oncology Associates, Augusta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - Hematology Oncology Centers of the Northern Rockies, Billings, Montana
  - Tri-County Oncology Hematology Associates, Canton, Ohio
  - Pacific Oncology, PC, Portland, Oregon
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Cancer Specialists of Tidewater, Chesapeake, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 community oncology research sites across the US within the ACORN network participated in this study. Enrollment started in August 2007 and was completed in September 2009.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent screening procedures to verify eligibility.
Groups:
- Pemetrexed, Gemcitabine, and Bevacizumab: All subjects received treatment with pemetrexed 500 mg/m^2, gemcitabine 1500 mg/m^2, and bevacizumab 10 mg/kg every 2 weeks.
Period: Overall Study
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 72.60 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first. Progression is defined per RECIST criteria v1.0 as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions. The median progression free survival is the parameter used to describe PFS.
Time Frame: PFS was measured from day 1 of treatment until time of progression (assessed every 8 weeks) or death, whichever came first, assessed up to 15 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Months | 4.90 [3.82 to 5.76]

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from treatment start until objective tumor progression. Progression is defined per RECIST criteria v1.0 as a measurable increase in the smallest diameter of any target lesion, progression of existing non-target lesions, or the appearance of 1 or more new lesions. The median time to progression is the parameter used to describe TTP.
Time Frame: TTP was measured from day 1 of treatment until time of progression (assessed every 8 weeks), assessed up to 15 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Months | 5.56 [4.61 to 7.57]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death from any cause. The median overall survival time is used to measure OS.
Time Frame: OS was measured from day 1 of treatment until time of death, assessed up to 20 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Months | 8.78 [6.71 to 19.9]

4. Secondary Outcome: Overall Response
Description: Response was evaluated via changes from baseline in radiological tumor measurements performed after every 4th treatment cycle and at the end of treatment or time of progression. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD) is neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD) is the increase in existing lesions or new lesions.
Time Frame: Response to treatment was assessed after every 8 weeks of treatment, up to 50 weeks.
Measure: Number; unit: Participants
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Participants
  Complete response (CR) | 0
  Partial response (PR) | 17
  Stable disease (SD) | 21
  Progressive disease (PD) | 6
  Not evaluable (NE) | 4

5. Other Pre Specified Outcome: Progression Free Survival (PFS) by Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first. The median progression free survival is the parameter used to describe PFS. ECOG performance status describes how daily living activities of the patient are affected by disease. ECOG of 0 means the patient is fully active without restriction. ECOG of 1 means the patient is restricted in physically strenuous activity but is able to carry out light work. The investigator assigned the ECOG score at baseline (i.e., before the patient started study treatment).
Time Frame: as for outcome 1
Population: Note that N=18 patients for the Baseline ECOG performance status 0 group, and N=30 patients for the Baseline ECOG performance status 1 group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Months
  Baseline ECOG performance status 0 (N=18) | 7.57 [2.01 to 9.44]
  Baseline ECOG performance status 1 (N=30) | 4.67 [3.68 to 5.30]
Statistical Analysis 1: Comparison: Pemetrexed, Gemcitabine, and Bevacizumab; Within Group 1 (N=48), patients with an ECOG of 0 at baseline (N=18) were compared to patients with an ECOG of 1 at baseline (N=30); Test type: Superiority or Other; p = 0.02, Log Rank

6. Other Pre Specified Outcome: Overall Survival (OS) by Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Overall survival is defined as the time from treatment start until death from any cause. The median overall survival time is used to measure OS. ECOG performance status describes how daily living activities of the patient are affected by disease. ECOG of 0 means the patient is fully active without restriction. ECOG of 1 means the patient is restricted in physically strenuous activity but is able to carry out light work. The investigator assigned the ECOG score at baseline (i.e., before the patient started study treatment).
Time Frame: OS was measured from day 1 of treatment until time of death, assessed up to 20 months.
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Number analyzed (Participants) | 48
Months
  Baseline ECOG performance status 0 (N=18) | 19.87 [4.90 to 19.9]
  Baseline ECOG performance status 1 (N=30) | 6.71 [4.67 to 8.78]
Statistical Analysis 1: Comparison: Pemetrexed, Gemcitabine, and Bevacizumab; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0041, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment, up to 54 weeks.
Arm/Group | Pemetrexed, Gemcitabine, and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 26/48
Other Adverse Events (participants affected / at risk) | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed, Gemcitabine, and Bevacizumab (N=48)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Adverse drug reaction (General disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 2
Edema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Hip fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed, Gemcitabine, and Bevacizumab (N=48)
Anemia (Blood and lymphatic system disorders) | 16
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Hypothyroidism (Endocrine disorders) | 1
Eye irritation (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 5
Periorbital edema (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Visual impairment (Eye disorders) | 1
Vitreous hemorrhage (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 15
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 18
Esophagitis (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 7
Catheter site erosion (General disorders) | 1
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 3
Device occlusion (General disorders) | 1
Face edema (General disorders) | 1
Fatigue (General disorders) | 30
Gait disturbance (General disorders) | 1
Irritability (General disorders) | 1
Malaise (General disorders) | 3
Mucosal inflammation (General disorders) | 5
Edema (General disorders) | 3
Edema peripheral (General disorders) | 9
Pain (General disorders) | 1
Pyrexia (General disorders) | 8
Swelling (General disorders) | 1
Thirst (General disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Anal abscess (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 3
Fungal infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localized infection (Infections and infestations) | 2
Lower respiratory infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 5
Skin infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 6
Vulvovaginal mycotic infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 1
Periorbital hematoma (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Glomerular filtration rate (Investigations) | 1
Neutrophil count (Investigations) | 2
Neutrophil count increased (Investigations) | 1
Occult blood positive (Investigations) | 1
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 7
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Cerebral atrophy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 4
Hypoesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Disorientation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 9
Mood altered (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Incontinence (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 6
Renal pain (Renal and urinary disorders) | 1
Urinary bladder hemorrhage (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Urogenital hemorrhage (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 7
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Catheter placement (Surgical and medical procedures) | 1
Embolism venous (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the proposed publication or presentation must be submitted to the funders for review and comment two months prior to the presentation or submission for publication. An additional 60 day delay of presentation or publication may be requested by the funder.